CLINICAL TRIAL: NCT01104402
Title: Early Intervention in Cystic Fibrosis Exacerbation
Acronym: eICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Washington (Other); National Institutes of Health (NIH) (NIH); Cystic Fibrosis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL001; LECHTZ10A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation); R01HL103965 (NIH)
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
Keywords: telemedicine; spirometer; CF; pulmonary; home monitoring
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Subjects will receive education about signs and symptoms indicative of worsening CF.
- Home monitoring (Active Comparator): Subjects will be randomized to monitor home spirometry and symptoms using a handheld device.
  Interventions: Device: Home lung function and symptom monitoring

INTERVENTIONS:
Device: Home lung function and symptom monitoring — subjects in the intervention arm will measure spirometry and CF symptoms with the use of a handheld device.
  Other Names: Jaeger AM2 monitor
  Arms: Home monitoring

SUMMARY:
Individuals with cystic fibrosis (CF) develop chronic lung infections and suffer intermittent acute exacerbations of their lung disease. Most exacerbations are not treated until they cause increased symptoms, and patients seek medical attention. This proposal details a study of home lung function and symptom monitoring. Subjects will be randomly assigned to one of two groups: 1) home monitoring, in which spirometry and symptoms are recorded; or 2) standard care. The home monitoring data will be transmitted electronically to the study center. If spirometry or symptoms have deteriorated substantially, treatment for a CF pulmonary exacerbation will be initiated. It is anticipated that use of home monitoring will lead to earlier, more reliable recognition and treatment of exacerbations, which will translate into better lung health.

DETAILED DESCRIPTION:
Individuals with CF develop chronic lung infections and suffer intermittent exacerbations, which require intensive treatment with antibiotics. The most common and useful objective measure of CF lung disease is spirometry. Chronic treatment of CF lung disease requires airway clearance, mucolytics and antibiotics. These treatments have been quite successful and there is evidence that early, aggressive treatment of lung disease results in better outcomes. Unfortunately, most exacerbations are not treated until they cause pronounced deterioration in symptoms, which prompts patients to seek medical attention. Self-monitoring of clinical status has improved outcomes in many other disorders such as asthma, diabetes mellitus, and lung transplantation. This is an important, randomized trial of home lung function and symptom monitoring in CF. Subjects will be assigned to one of two groups: 1) Home monitoring, in which spirometry and symptoms are recorded daily; or 2) Standard Care. The home monitoring data will be transmitted electronically twice weekly to the study center, where the results will be reviewed. If spirometry or symptoms have deteriorated substantially below baseline, treatment for a CF pulmonary exacerbation will be initiated. It is anticipated that use of home monitoring will translate into better clinical outcomes. We will test the hypothesis that if pulmonary exacerbations are identified and treated earlier than the current standard of care, the progression of lung disease will be slowed.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosis confirmed with sweat test, abnormal nasal potential difference and/or genetic testing
* Age 14 and older
* Able to perform spirometry
* Clinically stable without antibiotic treatment for a pulmonary exacerbation in the two weeks prior to the screening visit
* Forced expiratory volume in the first second (FEV1) greater than 25% of predicted at screening

Exclusion Criteria:

* History of solid organ transplant
* Participation in any interventional trial within the last 30 days
* Inability to speak and read the English language well enough to complete questionnaires
* Colonization with Burkholderia cepacia genomovar III within the last 24 months
* Currently receiving antimicrobial treatment specifically used to treat active non-tuberculosis mycobacterium
* Confirmed diagnosis of allergic bronchopulmonary aspergillosis (ABPA) as defined by the Cystic Fibrosis Foundation (CFF) guidance document that is being actively treated

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lechtzin, MD, Principal Investigator — Johns Hopkins University; Christopher Goss, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Johns Hopkins University CF Clinic, Baltimore, Maryland
  - University of Washington, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] VanDevanter EJ, Heltshe SL, Skalland M, Lechtzin N, Nichols D, Goss CH. The effect of oral and intravenous antimicrobials on pulmonary exacerbation recovery in cystic fibrosis. J Cyst Fibros. 2021 Nov;20(6):932-936. doi: 10.1016/j.jcf.2021.02.012. Epub 2021 Mar 5. PMID 33685776
- [Derived] Lechtzin N, Mayer-Hamblett N, West NE, Allgood S, Wilhelm E, Khan U, Aitken ML, Ramsey BW, Boyle MP, Mogayzel PJ Jr, Gibson RL, Orenstein D, Milla C, Clancy JP, Antony V, Goss CH; eICE Study Team. Home Monitoring of Patients with Cystic Fibrosis to Identify and Treat Acute Pulmonary Exacerbations. eICE Study Results. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1144-1151. doi: 10.1164/rccm.201610-2172OC. PMID 28608719

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Home Monitoring
Started | 132 | 135
Completed | 111 | 102
Not Completed | 21 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Home Monitoring | Total
Number analyzed (Participants) | 132 | 135 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 38 | 77
  Between 18 and 65 years | 93 | 97 | 190
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (12.5) | 26.5 (11.5) | 27.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 68 | 136
  Male | 64 | 67 | 131
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 132 | 135 | 267

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1
Description: The primary outcome variable is FEV1 which will be obtained at quarterly study visits. The primary analysis will use a linear mixed effects model incorporating all FEV1 measurements to estimate the 52-week change in FEV1
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
Liters | -0.07 [-.13 to -.02] | -0.08 [-.13 to -.03]

2. Secondary Outcome: Cystic Fibrosis Respiratory Symptom Diary (CFRSD)
Description: Change in CF respiratory symptoms as measured by the CFRSD. The CFRSD consists of 8 items which quantify symptom severity for the previous 24 hours to capture the magnitude of symptoms in stable CF, during medically treated CF exacerbations, and during recovery from an exacerbation. The CFRSD also includes emotional and activity impacts. Emotional impacts include frustration, sadness/depression, irritability, worry, and difficulty sleeping. Activity impacts include time spent sitting or lying down, reduction of usual activities, and missing school or work. will be analyzed using a linear mixed effects model incorporating baseline randomization factors FEV1 (<50%, 50-75%, and >75% predicted) and age (14-18 & 19+), treatment group, time (in weeks) and the interaction between treatment and time. The range of scores is 8 to 40 with higher scores indicating more severe symptoms.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
units on a scale | 4.56 (12.8) | 0.45 (13.6)

3. Secondary Outcome: Pulmonary Exacerbations
Description: Percentage of participants who experienced at least one acute pulmonary exacerbation
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
percentage of participants | 70 | 75

4. Secondary Outcome: Change in Health Related Quality of Life Scores as Assessed by the Cystic Fibrosis Questionnaire Revised (CFQ-R) (Respiratory Subscale Only(
Description: Change in health related quality of life as measured by the Cystic Fibrosis Questionnaire revised (CFQ-R)will be analyzed using a linear mixed effects model incorporating baseline randomization factors FEV1 (<50%, 50-75%, and >75% predicted) and age (14-18 & 19+), treatment group, time (in weeks) and the interaction between treatment and time. The CFQ-R measures functioning in a variety of domains, including Physical Functioning, Vitality, Health Perceptions, Respiratory Symptoms, Treatment Burden, Role Functioning, Emotional Functioning, and Social Functioning. Only the respiratory subscale of the the CFQ-R was evaluated. This ranges from 0 to 100 with higher scores indicating better respiratory quality of life. A negative number indicates a decrease in respiratory quality of life.
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
units on a scale | -3.07 (15.5) | -.44 (16.67)

5. Secondary Outcome: Treatment Burden
Description: Change in treatment burden as measured by the Cystic Fibrosis Questionnaire revised (CFQ-R)will be analyzed using a linear mixed effects model incorporating baseline randomization factors FEV1 (<50%, 50-75%, and >75% predicted) and age (14-18 & 19+), treatment group, time (in weeks) and the interaction between treatment and time. Scores range from 0-100 with higher scores indicating less treatment burden.
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 111 | 102
units on a scale | 0.6 (1.4) | 2.9 (2.6)

6. Secondary Outcome: Change in Prevalence of Resistant Species of Bacteria
Description: Change in prevalence of resistant species of bacteria (Methicillin Resistant S. aureus, Pseudomonas aeruginosa, Burkolderia cepacia, Stenotrophomona maltophilia, Achromobacterxylosoxidans) in sputum between baseline and final visit (Visit 5 or early withdrawal) will be summarized by treatment group.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects with new MRPA
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
percentage of subjects with new MRPA | 3 | 8

7. Secondary Outcome: Serious Adverse Events (SAE)
Description: Adverse event rates will be coded by body system and MedDRA classification term. Adverse events will be tabulated by treatment group and will include the number of subjects for whom the event occurred, the rate of occurrence, and the severity and relationship to study participation or study procedures.
Time Frame: 12 months
Measure: Number; unit: proportion of participants with SAEs
Arm/Group | Standard Care | Home Monitoring
Number analyzed (Participants) | 132 | 135
proportion of participants with SAEs | 0.023 | 0.030

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Care | Home Monitoring
Serious Adverse Events (participants affected / at risk) | 3/132 | 4/135
Other Adverse Events (participants affected / at risk) | 47/132 | 53/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=132) | Home Monitoring (N=135)
Exacerbation of Cystic Fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=132) | Home Monitoring (N=135)
nausea (Gastrointestinal disorders) | 10 (10) | 16 (17)
sputum increased (Respiratory, thoracic and mediastinal disorders) | 37 (153) | 37 (187)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No